CLINICAL TRIAL: NCT00696657
Title: Investigation of Safety and Efficacy of Five Doses of Semaglutide Versus Placebo and Open-label Liraglutide, as Add on Therapy, in Subjects Diagnosed With Type 2 Diabetes Currently Treated With Metformin or Controlled With Diet and Exercise A 12 Week Multi-centre, Multi National, Double-blind, Placebo-controlled, Randomised, Nine Armed Parallel Group, Dose Finding Trial
Brief Title: A Randomised Controlled Clinical Trial in Type 2 Diabetes Comparing Semaglutide to Placebo and Liraglutide
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9535-1821; 2007-003956-12 (EudraCT Number)
Record Dates: First submitted 2008-06-11; First posted 2008-06-13 (Estimated); Results first posted 2018-09-12 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-07

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — semaglutide; Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (14):
- A (Experimental)
  Interventions: Drug: semaglutide
- B (Experimental)
  Interventions: Drug: semaglutide
- C (Experimental)
  Interventions: Drug: semaglutide
- D (Experimental)
  Interventions: Drug: semaglutide
- E (Experimental)
  Interventions: Drug: semaglutide
- F (Experimental)
  Interventions: Drug: semaglutide
- G1 (Placebo Comparator)
  Interventions: Drug: placebo
- G2 (Placebo Comparator)
  Interventions: Drug: placebo
- G3 (Placebo Comparator)
  Interventions: Drug: placebo
- G4 (Placebo Comparator)
  Interventions: Drug: placebo
- G5 (Placebo Comparator)
  Interventions: Drug: placebo
- G6 (Placebo Comparator)
  Interventions: Drug: placebo
- H (Experimental)
  Interventions: Drug: liraglutide
- I (Experimental)
  Interventions: Drug: liraglutide

INTERVENTIONS:
Drug: semaglutide — 0.1 mg, once weekly, s.c. injection
  Other Names: NN9535
  Arms: A
Drug: semaglutide — 0.2 mg, once weekly, s.c. injection
  Other Names: NN9535
  Arms: B
Drug: semaglutide — 0.4 mg, once weekly, s.c. injection
  Other Names: NN9535
  Arms: C
Drug: semaglutide — 0.8 mg, once weekly, s.c. injection
  Other Names: NN9535
  Arms: D
Drug: semaglutide — 0.8 mg with titration, once weekly, s.c. injection
  Other Names: NN9535
  Arms: E
Drug: semaglutide — 1.6 mg with titration, once weekly, s.c. injection
  Other Names: NN9535
  Arms: F
Drug: placebo — 0.1 mg, once weekly, s.c. injection
  Arms: G1
Drug: placebo — 0.2 mg, once weekly, s.c. injection
  Arms: G2
Drug: placebo — 0.4 mg, once weekly, s.c. injection
  Arms: G3
Drug: placebo — 0.8 mg with titration, once weekly, s.c. injection
  Arms: G4; G5
Drug: placebo — 1.6 mg, once weekly, s.c. injection
  Arms: G6
Drug: liraglutide — 1.2 mg with titration, once daily, s.c. injection
  Arms: H
Drug: liraglutide — 1.8 mg with titration, once daily, s.c. injection
  Arms: I

SUMMARY:
This trial was conducted in Europe,Asia and Africa. Study participants were randomised evenly to treatment with semaglutide (0.1 mg QW - 1.6 mg QW, 6 treatment arms, placebo or liraglutide (1.2 mg QD, or 1.8 mg QD).Treatment allocation to semaglutide or placebo was double-blind, whereas liraglutide treatment was administered open-label.Primary efficacy parameter was HbA1c and the treatment duration was 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Men and women-not-of-childbearing potential diagnosed with type 2 diabetes for at least three months
* Stable treatment regimen with either metformin (at least 1500 mg) or diet and exercise alone for at least three months
* HbA1c: 7.0-10.0 % (both inclusive)
* Body weight between 60 kg and 110 kg

Exclusion Criteria:

* Treatment with insulin, GLP-1 receptor agonists (including liraglutide), dipeptidyl peptidase-4 inhibitors, sulphonylurea, thiazolidinediones, Alpha-GIs, or any investigational drug, within the last three months
* Impaired liver or kidney function
* Proliferative retinopathy or maculopathy requiring acute treatment
* Clinically significant active cardiovascular disease and uncontrolled treated/untreated hypertension
* Recurrent major hypoglycaemia or hypoglycaemic unawareness
* Present or planned use of any drug which could interfere with the glucose levels (e.g. systemic corticosteroids)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 415 (Actual)
Dates: Start 2008-06-03 (Actual); Primary Completion 2009-02-05 (Actual); Study Completion 2009-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry B. (GCR, 1452), MD, PhD, Study Director — Novo Nordisk A/S
Locations (68):
- Austria (5):
  - Novo Nordisk Investigational Site, Gratwein
  - Novo Nordisk Investigational Site, Graz
  - Novo Nordisk Investigational Site, Innsbruck
  - Novo Nordisk Investigational Site, Mödling
  - Novo Nordisk Investigational Site, Vienna
- Bulgaria (4):
  - Novo Nordisk Investigational Site, Plovdiv
  - Novo Nordisk Investigational Site, Rousse
  - Novo Nordisk Investigational Site, Sofia
  - Novo Nordisk Investigational Site, Varna
- Finland (6):
  - Novo Nordisk Investigational Site, Helsinki
  - Novo Nordisk Investigational Site, Imatra
  - Novo Nordisk Investigational Site, Mikkeli
  - Novo Nordisk Investigational Site, Oulu
  - Novo Nordisk Investigational Site, Tampere
  - Novo Nordisk Investigational Site, Turku
- France (5):
  - Novo Nordisk Investigational Site, Dommartin-lès-Toul
  - Novo Nordisk Investigational Site, La Rochelle
  - Novo Nordisk Investigational Site, Montpellier
  - Novo Nordisk Investigational Site, Narbonne
  - Novo Nordisk Investigational Site, Vénissieux
- Germany (7):
  - Novo Nordisk Investigational Site, Bad Lauterberg im Harz
  - Novo Nordisk Investigational Site, Falkensee
  - Novo Nordisk Investigational Site, Hamburg
  - Novo Nordisk Investigational Site, Ludwigshafen
  - Novo Nordisk Investigational Site, Marburg
  - Novo Nordisk Investigational Site, Münster
  - Novo Nordisk Investigational Site, Pohlheim
- Hungary (5):
  - Novo Nordisk Investigational Site, Budapest
  - Novo Nordisk Investigational Site, Debrecen
  - Novo Nordisk Investigational Site, Gyula
  - Novo Nordisk Investigational Site, Pécs
  - Novo Nordisk Investigational Site, Szekszárd
- India (4):
  - Novo Nordisk Investigational Site, Hyderabad, Andhra Pradesh
  - Novo Nordisk Investigational Site, Chennai, Tamil Nadu
  - Novo Nordisk Investigational Site, Chennai
  - Novo Nordisk Investigational Site, Hyderabad
- Italy (6):
  - Novo Nordisk Investigational Site, Catanzaro
  - Novo Nordisk Investigational Site, Chieti
  - Novo Nordisk Investigational Site, Florence
  - Novo Nordisk Investigational Site, Milano (MI)
  - Novo Nordisk Investigational Site, Napoli
  - Novo Nordisk Investigational Site, Perugia
- Novo Nordisk Investigational Site, Belgrade, Serbia and Montenegro
- South Africa (3):
  - Novo Nordisk Investigational Site, Pretoria, Gauteng
  - Novo Nordisk Investigational Site, Durban, KwaZulu-Natal
  - Novo Nordisk Investigational Site, Cape Town, Western Cape
- Spain (5):
  - Novo Nordisk Investigational Site, Almería
  - Novo Nordisk Investigational Site, Gijón
  - Novo Nordisk Investigational Site, Madrid
  - Novo Nordisk Investigational Site, Seville
  - Novo Nordisk Investigational Site, Valencia
- Switzerland (4):
  - Novo Nordisk Investigational Site, Bern
  - Novo Nordisk Investigational Site, Geneva
  - Novo Nordisk Investigational Site, Lausanne
  - Novo Nordisk Investigational Site, Sankt Gallen
- Turkey (Türkiye) (2):
  - Novo Nordisk Investigational Site, Antalya
  - Novo Nordisk Investigational Site, Istanbul
- United Kingdom (11):
  - Novo Nordisk Investigational Site, Addlestone
  - Novo Nordisk Investigational Site, Bath
  - Novo Nordisk Investigational Site, Bexhill-on-Sea
  - Novo Nordisk Investigational Site, Bradford
  - Novo Nordisk Investigational Site, Dundee
  - Novo Nordisk Investigational Site, Guildford
  - Novo Nordisk Investigational Site, Hull
  - Novo Nordisk Investigational Site, Inverness
  - Novo Nordisk Investigational Site, Llanelli
  - Novo Nordisk Investigational Site, Sheffield
  - Novo Nordisk Investigational Site, Trowbridge

REFERENCES:
- [Derived] Nauck MA, Petrie JR, Sesti G, Mannucci E, Courreges JP, Lindegaard ML, Jensen CB, Atkin SL; Study 1821 Investigators. A Phase 2, Randomized, Dose-Finding Study of the Novel Once-Weekly Human GLP-1 Analog, Semaglutide, Compared With Placebo and Open-Label Liraglutide in Patients With Type 2 Diabetes. Diabetes Care. 2016 Feb;39(2):231-41. doi: 10.2337/dc15-0165. Epub 2015 Sep 10. PMID 26358288
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 80 sites in 14 countries: Austria (8), Bulgaria (6), Finland (6), France (5), Germany (7), Hungary (5), India (4), Italy (6), Serbia (3), South Africa (3), Spain (6), Switzerland (4), Turkey (5), and United Kingdom (12).
Pre-assignment Details: Study Design: This was a 9 armed parallel group trial. Subjects were randomised in a 1:1:1:1:1:1:1:1:1 manner to receive one of five doses of blinded semaglutide once-weekly (0.1 mg, 0.2 mg, 0.4 mg, 0.8 mg, 0.8 mg T [with titration] and 1.6 mg T [with titration]) or blinded placebo once-weekly or open-label liraglutide 1.2 mg or 1.8 mg once-daily.
Groups:
- Placebo: Subjects received placebo once-weekly throughout the 12-week treatment period. Placebo was injected subcutaneously (s.c.; under the skin) in the abdomen, thigh or upper arm by using the NordiPen® on the same day of the week at a convenient time for the subjects. Placebo was given in adjunct to previous metformin therapy on a stable dose (minimum 1.5 g daily) or as monotherapy in case the diabetes was controlled by diet and exercise alone.
- Semaglutide 0.1 mg: Subjects received semaglutide 0.1 mg once-weekly throughout the 12-week treatment period. Semaglutide was injected s.c. in the abdomen, thigh or upper arm by using the NordiPen® on the same day of the week at a convenient time for the subjects. Semaglutide was given in adjunct to previous metformin therapy on a stable dose (minimum 1.5 g daily) or as monotherapy in case the diabetes was controlled by diet and exercise alone.
- Semaglutide 0.2 mg: Subjects received semaglutide 0.2 mg once-weekly throughout the 12-week treatment period. Semaglutide was injected s.c. in the abdomen, thigh or upper arm by using the NordiPen® on the same day of the week at a convenient time for the subjects. Semaglutide was given in adjunct to previous metformin therapy on a stable dose (minimum 1.5 g daily) or as monotherapy in case the diabetes was controlled by diet and exercise alone.
- Semaglutide 0.4 mg: Subjects received semaglutide 0.4 mg once-weekly throughout the 12-week treatment period. Semaglutide was injected s.c. in the abdomen, thigh or upper arm by using the NordiPen® on the same day of the week at a convenient time for the subjects. Semaglutide was given in adjunct to previous metformin therapy on a stable dose (minimum 1.5 g daily) or as monotherapy in case the diabetes was controlled by diet and exercise alone.
- Semaglutide 0.8 mg: Subjects received semaglutide 0.8 mg once-weekly throughout the 12-week treatment period. Semaglutide was injected s.c. in the abdomen, thigh or upper arm by using the NordiPen® on the same day of the week at a convenient time for the subjects. Semaglutide was given in adjunct to previous metformin therapy on a stable dose (minimum 1.5 g daily) or as monotherapy in case the diabetes was controlled by diet and exercise alone.
- Semaglutide 0.8 mg (With Titration): Subjects followed a 1-week titration period (semaglutide 0.4 mg once-weekly at week 1), followed by an 11- week treatment period of fixed doses semaglutide 0.8 mg, once-weekly. Semaglutide was injected s.c. in the abdomen, thigh or upper arm by using the NordiPen® on the same day of the week at a convenient time for the subjects. Semaglutide was given in adjunct to previous metformin therapy on a stable dose (minimum 1.5 g daily) or as monotherapy in case the diabetes was controlled by diet and exercise alone.
- Semaglutide 1.6 mg (With Titration): Subjects followed a 2-week titration period (once-weekly semaglutide 0.4 mg at week 1 and 0.8 mg at week 2), followed by a 10-week treatment period of fixed doses semaglutide 1.6 mg, once-weekly. Semaglutide was injected s.c. in the abdomen, thigh or upper arm by using the NordiPen® on the same day of the week at a convenient time for the subjects. Semaglutide was given in adjunct to previous metformin therapy on a stable dose (minimum 1.5 g daily) or as monotherapy in case the diabetes was controlled by diet and exercise alone.
- Liraglutide 1.2 mg: Subjects followed a 1-week titration period (liraglutide 0.6 mg once-daily in week 1), followed by an 11-week treatment period of fixed doses liraglutide 1.2 mg, once-daily. Liraglutide was injected s.c. in the abdomen, upper arm or thigh by using the Flexpen® in the evening before bedtime. Liraglutide was given in adjunct to previous metformin therapy on a stable dose (minimum 1.5 g daily) or as monotherapy in case the diabetes was controlled by diet and exercise alone.
- Liraglutide 1.8 mg: Subjects followed a 2-week titration period (once-daily liraglutide 0.6 mg in week 1 and 1.2 mg in week 2), followed by a 10-week treatment period of fixed doses liraglutide 1.8 mg, once-daily. Liraglutide was injected s.c. in the abdomen, upper arm or thigh by using the Flexpen® in the evening before bedtime. Liraglutide was given in adjunct to previous metformin therapy on a stable dose (minimum 1.5 g daily) or as monotherapy in case the diabetes was controlled by diet and exercise alone.
Period: Overall Study
Arm/Group | Placebo | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Semaglutide 0.8 mg | Semaglutide 0.8 mg (With Titration) | Semaglutide 1.6 mg (With Titration) | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Started (STARTED = Randomised.) | 46 | 47 | 44 | 49 | 44 | 45 | 45 | 45 | 50
EXPOSED | 46 | 47 | 43 | 48 | 44 | 43 | 45 | 45 | 50
Completed | 45 | 42 | 36 | 38 | 34 | 33 | 30 | 42 | 41
Not Completed | 1 | 5 | 8 | 11 | 10 | 12 | 15 | 3 | 9
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal criteria | 1 | 3 | 2 | 2 | 0 | 0 | 1 | 1 | 2
Not completed — Unclassified | 0 | 1 | 3 | 2 | 4 | 2 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 3 | 7 | 6 | 9 | 14 | 2 | 5

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all randomised subjects who were exposed to at least 1 dose of trial product. 2 subjects randomised to semaglutide 0.8mg were mistakenly titrated, so actual treatment was semaglutide 0.8mg T. 2 subjects randomised to semaglutide 0.8mg T were mistakenly titrated to 1.6mg T, so actual treatment was semaglutide 1.6mg T
Groups:
- Placebo: Subjects received placebo once-weekly throughout the 12-week treatment period. Placebo was injected s.c. in the abdomen, thigh or upper arm by using the NordiPen® on the same day of the week at a convenient time for the subjects. Placebo was given in adjunct to previous metformin therapy on a stable dose (minimum 1.5 g daily) or as monotherapy in case the diabetes was controlled by diet and exercise alone.
- Total: Total of all reporting groups
Arm/Group | Placebo | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Semaglutide 0.8 mg | Semaglutide 0.8 mg (With Titration) | Semaglutide 1.6 mg (With Titration) | Liraglutide 1.2 mg | Liraglutide 1.8 mg | Total
Number analyzed (Participants) | 46 | 47 | 43 | 48 | 42 | 43 | 47 | 45 | 50 | 411
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.3 (10.6) | 55.2 (10.1) | 54.7 (10.0) | 53.8 (10.2) | 55.0 (9.7) | 55.9 (7.9) | 56.4 (10.5) | 54.8 (9.2) | 54.3 (10.1) | 55.0 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 16 | 13 | 11 | 20 | 16 | 21 | 14 | 15 | 144
  Male | 28 | 31 | 30 | 37 | 22 | 27 | 26 | 31 | 35 | 267
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: Percentage (%) of HbA1c] | 8.1 (0.8) | 8.2 (0.9) | 8.2 (0.9) | 8.1 (0.9) | 8.2 (0.9) | 8.0 (0.8) | 8.0 (0.7) | 8.0 (0.8) | 8.1 (0.7) | 8.1 (0.8)
Systolic blood pressure (SBP) [Mean (Standard Deviation); unit: mmHg] | 130.9 (13.1) | 129.4 (11.6) | 129.3 (13.4) | 134.0 (12.9) | 132.6 (13.3) | 130.3 (13.0) | 131.1 (10.7) | 128.0 (10.2) | 130.4 (13.9) | 130.7 (12.5)
Diastolic blood pressure (DBP) [Mean (Standard Deviation); unit: mmHg] | 79.1 (8.3) | 79.1 (6.5) | 79.3 (7.6) | 81.9 (7.5) | 80.8 (7.9) | 79.4 (9.3) | 80.9 (8.9) | 80.0 (9.2) | 78.9 (7.7) | 79.9 (8.1)
Pulse [Mean (Standard Deviation); unit: Beats/min] | 70.4 (9.2) | 74.2 (8.0) | 72.8 (9.0) | 74.3 (9.2) | 74.7 (8.7) | 74.2 (10.2) | 73.9 (9.7) | 72.3 (7.5) | 74.6 (10.8) | 73.5 (9.2)

OUTCOME MEASURES:

1. Primary Outcome: HbA1c
Description: Change from baseline in HbA1c was evaluated after 12 weeks of treatment. Post baseline (week 0) missing values were replaced using the last observation carried forward (LOCF) approach.
Time Frame: After 12 weeks of treatment.
Population: The full analysis set included all randomised subjects who had been exposed to at least 1 dose of the trial product (placebo/semaglutide/liraglutide). Four subjects mistakenly received a different treatment instead of the randomised treatment. The randomised treatment was applied regardless of the treatment actually received.
Measure: Mean (Standard Deviation); unit: Percentage (%) of HbA1c
Arm/Group | Placebo | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Semaglutide 0.8 mg | Semaglutide 0.8 mg (With Titration) | Semaglutide 1.6 mg (With Titration) | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 47 | 43 | 48 | 44 | 43 | 45 | 45 | 50
Percentage (%) of HbA1c | -0.5 (0.8) | -0.6 (0.7) | -0.9 (0.9) | -1.0 (0.8) | -1.4 (0.8) | -1.4 (1.0) | -1.5 (0.8) | -1.1 (0.7) | -1.3 (0.7)
Statistical Analysis 1: Comparison: Placebo vs Semaglutide 1.6 mg (With Titration); The comparison sequence should be read as "Semaglutide 1.6 mg (with titration) - Placebo". The estimates are from an analysis of variance (ANOVA) model with treatment, country and previous treatment as fixed effects and baseline HbA1c as covariate; Test type: Superiority; p < 0.0001, ANOVA; Confidence interval (CIs) for treatment differences versus placebo are based on Dunnett's method; Estimated treatment differences = -1.19, 95% CI 2-sided [-1.58 to -0.80]
Statistical Analysis 2: Comparison: Placebo vs Semaglutide 0.8 mg (With Titration); The comparison sequence should be read as "Semaglutide 0.8 mg (with titration) - Placebo". The estimates are from an ANOVA model with treatment, country and previous treatment as fixed effects and baseline HbA1c as covariate; Test type: Superiority; p < 0.0001, ANOVA; CIs for treatment differences versus placebo are based on Dunnett's method; Estimated treatment differences = -0.95, 95% CI 2-sided [-1.33 to -0.57]
Statistical Analysis 3: Comparison: Placebo vs Semaglutide 0.8 mg; The comparison sequence should be read as "Semaglutide 0.8 mg - Placebo". The estimates are from an ANOVA model with treatment, country and previous treatment as fixed effects and baseline HbA1c as covariate; Test type: Superiority; p < 0.0001, ANOVA; CIs for treatment differences versus placebo are based on Dunnett's method; Estimated treatment differences = -0.97, 95% CI 2-sided [-1.35 to -0.59]
Statistical Analysis 4: Comparison: Placebo vs Semaglutide 0.4 mg; The comparison sequence should be read as "Semaglutide 0.4 mg - Placebo". The estimates are from an ANOVA model with treatment, country and previous treatment as fixed effects and baseline HbA1c as covariate; Test type: Superiority; p = 0.0002, ANOVA; CIs for treatment differences versus placebo are based on Dunnett's method; Estimated treatment differences = -0.61, 95% CI 2-sided [-0.98 to -0.23]
Statistical Analysis 5: Comparison: Placebo vs Semaglutide 0.2 mg; The comparison sequence should be read as "Semaglutide 0.2 mg - Placebo". The estimates are from an ANOVA model with treatment, country and previous treatment as fixed effects and baseline HbA1c as covariate; Test type: Superiority; p = 0.0324, ANOVA; CIs for treatment differences versus placebo are based on Dunnett's method; Estimated treatment differences = -0.41, 95% CI 2-sided [-0.79 to -0.02]
Statistical Analysis 6: Comparison: Placebo vs Semaglutide 0.1 mg; The comparison sequence should be read as "Semaglutide 0.1 mg - Placebo". The estimates are from an ANOVA model with treatment, country and previous treatment as fixed effects and baseline HbA1c as covariate; Test type: Superiority; p = 0.9772, ANOVA; CIs for treatment differences versus placebo are based on Dunnett's method; Estimated treatment differences = -0.09, 95% CI 2-sided [-0.46 to 0.28]
Statistical Analysis 7: Comparison: Semaglutide 1.6 mg (With Titration) vs Liraglutide 1.8 mg; The comparison sequence should be read as "Semaglutide 1.6 mg (with titration) - Liraglutide 1.8 mg". The estimates are from an ANOVA model with treatment, country and previous treatment as fixed effects and baseline HbA1c as covariate; Test type: Other; ANOVA; CIs for treatment differences versus liraglutide are not corrected for multiple testing; Estimated treatment differences = -0.35, 95% CI 2-sided [-0.64 to -0.06]
Statistical Analysis 8: Comparison: Semaglutide 0.8 mg (With Titration) vs Liraglutide 1.8 mg; The comparison sequence should be read as "Semaglutide 0.8 mg (with titration) - Liraglutide 1.8 mg". The estimates are from an ANOVA model with treatment, country and previous treatment as fixed effects and baseline HbA1c as covariate; Test type: Other; ANOVA; CIs for treatment differences versus liraglutide are not corrected for multiple testing; Estimated treatment differences = -0.11, 95% CI 2-sided [-0.39 to 0.18]
Statistical Analysis 9: Comparison: Semaglutide 0.8 mg vs Liraglutide 1.8 mg; The comparison sequence should be read as "Semaglutide 0.8 mg - Liraglutide 1.8 mg". The estimates are from an ANOVA model with treatment, country and previous treatment as fixed effects and baseline HbA1c as covariate; Test type: Other; ANOVA; CIs for treatment differences versus liraglutide are not corrected for multiple testing; Estimated treatment differences = -0.13, 95% CI 2-sided [-0.42 to 0.16]
Statistical Analysis 10: Comparison: Semaglutide 0.4 mg vs Liraglutide 1.8 mg; The comparison sequence should be read as "Semaglutide 0.4 mg - Liraglutide 1.8 mg". The estimates are from an ANOVA model with treatment, country and previous treatment as fixed effects and baseline HbA1c as covariate; Test type: Other; ANOVA; CIs for treatment differences versus liraglutide are not corrected for multiple testing; Estimated treatment differences = 0.24, 95% CI 2-sided [-0.05 to 0.52]
Statistical Analysis 11: Comparison: Semaglutide 0.2 mg vs Liraglutide 1.8 mg; The comparison sequence should be read as "Semaglutide 0.2 mg - Liraglutide 1.8 mg". The estimates are from an ANOVA model with treatment, country and previous treatment as fixed effects and baseline HbA1c as covariate; Test type: Other; ANOVA; CIs for treatment differences versus liraglutide are not corrected for multiple testing; Estimated treatment differences = 0.44, 95% CI 2-sided [0.15 to 0.73]
Statistical Analysis 12: Comparison: Semaglutide 0.1 mg vs Liraglutide 1.8 mg; The comparison sequence should be read as "Semaglutide 0.1 mg - Liraglutide 1.8 mg". The estimates are from an ANOVA model with treatment, country and previous treatment as fixed effects and baseline HbA1c as covariate; Test type: Other; ANOVA; CIs for treatment differences versus liraglutide are not corrected for multiple testing; Estimated treatment differences = 0.75, 95% CI 2-sided [0.48 to 1.03]
Statistical Analysis 13: Comparison: Placebo vs Liraglutide 1.8 mg; The comparison sequence should be read as "Liraglutide 1.8 mg - Placebo ". The estimates are from an ANOVA model with treatment, country and previous treatment as fixed effects and baseline HbA1c as covariate; Test type: Other; ANOVA; CIs for treatment differences versus liraglutide are not corrected for multiple testing; Estimated treatment differences = -0.84, 95% CI 2-sided [-1.12 to -0.56]
Statistical Analysis 14: Comparison: Semaglutide 1.6 mg (With Titration) vs Liraglutide 1.2 mg; The comparison sequence should be read as "Semaglutide 1.6 mg (with titration) - Liraglutide 1.2 mg". The estimates are from an ANOVA model with treatment, country and previous treatment as fixed effects and baseline HbA1c as covariate; Test type: Other; ANOVA; CIs for treatment differences versus liraglutide are not corrected for multiple testing; Estimated treatment differences = -0.51, 95% CI 2-sided [-0.80 to -0.22]
Statistical Analysis 15: Comparison: Semaglutide 0.8 mg (With Titration) vs Liraglutide 1.2 mg; The comparison sequence should be read as "Semaglutide 0.8 mg (with titration) - Liraglutide 1.2 mg". The estimates are from an ANOVA model with treatment, country and previous treatment as fixed effects and baseline HbA1c as covariate; Test type: Other; ANOVA; CIs for treatment differences versus liraglutide are not corrected for multiple testing; Estimated treatment differences = -0.27, 95% CI 2-sided [-0.56 to 0.02]
Statistical Analysis 16: Comparison: Semaglutide 0.8 mg vs Liraglutide 1.2 mg; The comparison sequence should be read as "Semaglutide 0.8 mg - Liraglutide 1.2 mg". The estimates are from an ANOVA model with treatment, country and previous treatment as fixed effects and baseline HbA1c as covariate; Test type: Other; ANOVA; CIs for treatment differences versus liraglutide are not corrected for multiple testing; Estimated treatment differences = -0.29, 95% CI 2-sided [-0.58 to 0.01]
Statistical Analysis 17: Comparison: Semaglutide 0.4 mg vs Liraglutide 1.2 mg; The comparison sequence should be read as "Semaglutide 0.4 mg - Liraglutide 1.2 mg". The estimates are from an ANOVA model with treatment, country and previous treatment as fixed effects and baseline HbA1c as covariate; Test type: Other; ANOVA; CIs for treatment differences versus liraglutide are not corrected for multiple testing; Estimated treatment differences = 0.08, 95% CI 2-sided [-0.22 to 0.37]
Statistical Analysis 18: Comparison: Semaglutide 0.2 mg vs Liraglutide 1.2 mg; The comparison sequence should be read as "Semaglutide 0.2 mg - Liraglutide 1.2 mg". The estimates are from an ANOVA model with treatment, country and previous treatment as fixed effects and baseline HbA1c as covariate; Test type: Other; ANOVA; CIs for treatment differences versus liraglutide are not corrected for multiple testing; Estimated treatment differences = 0.28, 95% CI 2-sided [-0.02 to 0.57]
Statistical Analysis 19: Comparison: Semaglutide 0.1 mg vs Liraglutide 1.2 mg; The comparison sequence should be read as "Semaglutide 0.1 mg - Liraglutide 1.2 mg". The estimates are from an ANOVA model with treatment, country and previous treatment as fixed effects and baseline HbA1c as covariate; Test type: Other; ANOVA; CIs for treatment differences versus liraglutide are not corrected for multiple testing; Estimated treatment differences = 0.59, 95% CI 2-sided [0.31 to 0.88]
Statistical Analysis 20: Comparison: Placebo vs Liraglutide 1.2 mg; The comparison sequence should be read as "Liraglutide 1.2 mg - Placebo". The estimates are from an ANOVA model with treatment, country and previous treatment as fixed effects and baseline HbA1c as covariate; Test type: Other; ANOVA; CIs for treatment differences versus liraglutide are not corrected for multiple testing; Estimated treatment differences = -0.68, 95% CI 2-sided [-0.97 to -0.40]

2. Secondary Outcome: Percentage of Subjects With an Adverse Events
Description: The results of adverse event presented here are treatment emergent, i.e., TEAE. A TEAE was defined as an event that had onset on or after the first date (week 0) on trial product and no later than 5 weeks after the last date on trial product (week 17), or that had onset before the first date on trial product and increases in severity during the treatment period until 5 weeks after the last date on trial product.
Time Frame: After 12 weeks of treatment.
Population: as for baseline characteristics
Measure: Number; unit: Percentage (%) of subjects
Arm/Group | Placebo | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Semaglutide 0.8 mg | Semaglutide 0.8 mg (With Titration) | Semaglutide 1.6 mg (With Titration) | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 47 | 43 | 48 | 42 | 43 | 47 | 45 | 45
Percentage (%) of subjects | 43.5 | 59.6 | 55.8 | 72.9 | 85.7 | 72.1 | 93.6 | 55.6 | 62.0

3. Secondary Outcome: Percentage of Subjects With Hypoglycaemic Episode
Description: The results of hypoglycaemic episode presented here are treatment emergent. Hypoglycaemic episodes were defined as treatment emergent if they had onset on or after the first day of randomised treatment (in week 0) and no later than 5 weeks after the last date on trial product (week 17). Hypoglycaemic episodes are classified as follows: Major: If the subject was not able to treat himself or herself and was needed to be administered food, glucagon or intravenous (i.v.) glucose by another person. Minor: If the subject was able to treat himself or herself and measured plasma glucose was <3.1 mmol/L (56 mg/dL). Symptoms only: If the subject was able to treat himself or herself and measured plasma glucose was >=3.1 mmol/L (56 mg/dL) or no plasma glucose measurement was done.
Time Frame: After 12 weeks of treatment
Population: as for baseline characteristics
Measure: Number; unit: Percentage (%) of subjects
Arm/Group | Placebo | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Semaglutide 0.8 mg | Semaglutide 0.8 mg (With Titration) | Semaglutide 1.6 mg (With Titration) | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 47 | 43 | 48 | 42 | 43 | 47 | 45 | 50
Percentage (%) of subjects
  Major | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Minor | 0 | 4.3 | 0 | 4.2 | 0 | 2.3 | 0 | 4.4 | 2.0
  Symptoms only | 2.2 | 2.1 | 2.3 | 0 | 0 | 0 | 6.4 | 8.9 | 2.0

4. Secondary Outcome: Change From Baseline in ECG
Description: A standard 12 lead electrocardiogram (ECG) with a 10-second rhythm strip was performed at screening (week -2) and at the end of treatment (week 12). The time frame should be read as "week -2, week 12". Change from baseline in ECG was measured in terms of number of subjects in each category (normal, abnormal, not clinically significant [NCS] or abnormal clinically significant [CS]) at week -2 and week 12 (i.e., change in each category in terms of number of subjects from week -2 to week 12).
Time Frame: Week 0, week 12.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Semaglutide 0.8 mg | Semaglutide 0.8 mg (With Titration) | Semaglutide 1.6 mg (With Titration) | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 47 | 43 | 48 | 42 | 43 | 47 | 45 | 50
Participants
  Week -2: Normal | 42 | 33 | 37 | 34 | 31 | 28 | 37 | 39 | 41
  Week -2: Abnormal, NCS | 4 | 14 | 6 | 12 | 10 | 15 | 8 | 6 | 9
  Week -2: Abnormal, CS | 0 | 0 | 0 | 2 | 1 | 0 | 2 | 0 | 0
  Week 12: Normal: number analyzed (Participants) | 46 | 47 | 43 | 46 | 40 | 43 | 46 | 45 | 49
  Week 12: Normal | 39 | 32 | 34 | 36 | 29 | 33 | 36 | 37 | 42
  Week 12: Abnormal, NCS: number analyzed (Participants) | 46 | 47 | 43 | 46 | 40 | 43 | 46 | 45 | 49
  Week 12: Abnormal, NCS | 6 | 14 | 3 | 7 | 7 | 9 | 5 | 6 | 5
  Week 12: Abnormal, CS: number analyzed (Participants) | 46 | 47 | 43 | 46 | 40 | 43 | 46 | 45 | 49
  Week 12: Abnormal, CS | 0 | 0 | 1 | 2 | 1 | 0 | 3 | 0 | 0
  Week 12: ECG not done (ND): number analyzed (Participants) | 46 | 47 | 43 | 46 | 40 | 43 | 46 | 45 | 49
  Week 12: ECG not done (ND) | 1 | 1 | 5 | 1 | 3 | 1 | 2 | 2 | 2

5. Secondary Outcome: Change From Baseline in Vital Signs (Pulse)
Description: Change from baseline in pulse was evaluated after 12 weeks of treatment. Post baseline (week 0) missing values were replaced using the LOCF approach.
Time Frame: Week 0, week 12
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Beats/minute
Arm/Group | Placebo | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Semaglutide 0.8 mg | Semaglutide 0.8 mg (With Titration) | Semaglutide 1.6 mg (With Titration) | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 47 | 43 | 48 | 42 | 43 | 47 | 45 | 50
Beats/minute | 0.5 (8.9) | -0.0 (7.6) | 0.5 (13.8) | 1.5 (8.5) | 1.5 (9.6) | 2.9 (11.9) | 3.9 (12.6) | 4.4 (10.2) | 2.1 (10.1)

6. Secondary Outcome: Change From Baseline in Vital Signs (Blood Pressure; SBP)
Description: Change from baseline in systolic blood pressure (SBP) was evaluated after 12 weeks of treatment. Post baseline (week 0) missing values were replaced using the LOCF approach.
Time Frame: Week 0, week 12
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Semaglutide 0.8 mg | Semaglutide 0.8 mg (With Titration) | Semaglutide 1.6 mg (With Titration) | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 47 | 43 | 48 | 42 | 43 | 47 | 45 | 50
mmHg | -3.2 (14.8) | 3.3 (11.0) | -2.5 (14.1) | -3.6 (13.1) | -6.7 (14.9) | -7.7 (13.0) | -5.9 (11.6) | -2.9 (12.0) | -5.4 (14.0)

7. Secondary Outcome: Change From Baseline in Vital Signs (Blood Pressure; DBP)
Description: Change from baseline in diastolic blood pressure (DBP) was evaluated after 12 weeks of treatment. Post baseline (week 0) missing values were replaced using the LOCF approach.
Time Frame: Week 0, week 12
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Semaglutide 0.8 mg | Semaglutide 0.8 mg (With Titration) | Semaglutide 1.6 mg (With Titration) | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 47 | 43 | 48 | 42 | 43 | 47 | 45 | 50
mmHg | -2.3 (9.8) | 1.5 (7.9) | -0.4 (8.5) | -1.5 (9.7) | -1.5 (7.9) | -2.3 (9.7) | -3.0 (7.7) | -2.1 (10.0) | -0.0 (8.8)

8. Secondary Outcome: Change From Baseline in Standard Safety Laboratory Parameter (Haematology; Basophils)
Description: Change from baseline in basophils was evaluated after 12 weeks of treatment. Post baseline (week 0) missing values were replaced using the LOCF approach.
Time Frame: Week 0, week 12
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Billion cells/litre (10^9/L)
Arm/Group | Placebo | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Semaglutide 0.8 mg | Semaglutide 0.8 mg (With Titration) | Semaglutide 1.6 mg (With Titration) | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 47 | 43 | 48 | 42 | 43 | 47 | 45 | 50
Billion cells/litre (10^9/L) | -0.0 (0.0) | 0.0 (0.0) | -0.0 (0.0) | 0.0 (0.0) | -0.0 (0.0) | -0.0 (0.0) | -0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)

9. Secondary Outcome: Change From Baseline in Standard Safety Laboratory Parameter (Haematology; Eosinophils)
Description: Change from baseline in eosinophils was evaluated after 12 weeks of treatment. Post baseline (week 0) missing values were replaced using the LOCF approach.
Time Frame: Week 0, week 12
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Billion cells/litre (10^9/L)
Arm/Group | Placebo | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Semaglutide 0.8 mg | Semaglutide 0.8 mg (With Titration) | Semaglutide 1.6 mg (With Titration) | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 47 | 43 | 48 | 42 | 43 | 47 | 45 | 50
Billion cells/litre (10^9/L) | -0.0 (0.2) | 0.0 (0.2) | -0.0 (0.1) | 0.0 (0.1) | -0.0 (0.2) | 0.0 (0.3) | 0.1 (0.2) | 0.0 (0.2) | -0.0 (0.1)

10. Secondary Outcome: Change From Baseline in Standard Safety Laboratory Parameter (Haematology; Haematocrit)
Description: Change from baseline in haematocrit (the proportion of blood that consists of red blood cells) was evaluated after 12 weeks of treatment. Post baseline (week 0) missing values were replaced using the LOCF approach.
Time Frame: Week 0, week 12
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Litre/litre (L/L)
Arm/Group | Placebo | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Semaglutide 0.8 mg | Semaglutide 0.8 mg (With Titration) | Semaglutide 1.6 mg (With Titration) | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 47 | 43 | 48 | 42 | 43 | 47 | 45 | 50
Litre/litre (L/L) | -0.01 (0.02) | -0.01 (0.03) | -0.01 (0.03) | 0.00 (0.03) | -0.01 (0.02) | -0.00 (0.03) | -0.00 (0.03) | 0.00 (0.03) | -0.01 (0.03)

11. Secondary Outcome: Change From Baseline in Standard Safety Laboratory Parameter (Haematology; Haemoglobin)
Description: Change from baseline in haemoglobin was evaluated after 12 weeks of treatment. Post baseline (week 0) missing values were replaced using the LOCF approach.
Time Frame: Week 0, week 12
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Gram/litre (g/L)
Arm/Group | Placebo | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Semaglutide 0.8 mg | Semaglutide 0.8 mg (With Titration) | Semaglutide 1.6 mg (With Titration) | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 47 | 43 | 48 | 42 | 43 | 47 | 45 | 50
Gram/litre (g/L) | 0.1 (6.3) | -0.4 (5.9) | -1.2 (9.3) | 2.8 (9.5) | -0.3 (7.7) | 1.5 (6.9) | 1.0 (7.1) | 2.1 (6.7) | 1.1 (10.7)

12. Secondary Outcome: Change From Baseline in Standard Safety Laboratory Parameter (Haematology; Lymphocytes)
Description: Change from baseline in lymphocytes was evaluated after 12 weeks of treatment. Post baseline (week 0) missing values were replaced using the LOCF approach.
Time Frame: Week 0, week 12
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Billion cells/litre (10^9/L)
Arm/Group | Placebo | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Semaglutide 0.8 mg | Semaglutide 0.8 mg (With Titration) | Semaglutide 1.6 mg (With Titration) | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 47 | 43 | 48 | 42 | 43 | 47 | 45 | 50
Billion cells/litre (10^9/L) | -0.1 (0.6) | 0.0 (0.4) | -0.1 (0.6) | 0.2 (0.9) | -0.0 (0.7) | -0.1 (0.7) | 0.1 (0.5) | 0.0 (0.4) | -0.1 (0.8)

13. Secondary Outcome: Change From Baseline in Standard Safety Laboratory Parameter (Haematology; Monocytes)
Description: Change from baseline in monocytes was evaluated after 12 weeks of treatment. Post baseline (week 0) missing values were replaced using the LOCF approach.
Time Frame: Week 0, week 12
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Billion cells/litre (10^9/L)
Arm/Group | Placebo | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Semaglutide 0.8 mg | Semaglutide 0.8 mg (With Titration) | Semaglutide 1.6 mg (With Titration) | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 47 | 43 | 48 | 42 | 43 | 47 | 45 | 50
Billion cells/litre (10^9/L) | 0.1 (0.1) | 0.0 (0.2) | -0.0 (0.2) | 0.1 (0.1) | 0.1 (0.2) | 0.0 (0.1) | 0.1 (0.2) | 0.1 (0.2) | 0.1 (0.2)

14. Secondary Outcome: Change From Baseline in Standard Safety Laboratory Parameter (Haematology; Neutrophils)
Description: Change from baseline in neutrophils was evaluated after 12 weeks of treatment. Post baseline (week 0) missing values were replaced using the LOCF approach.
Time Frame: Week 0, week 12
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Billion cells/litre (10^9/L)
Arm/Group | Placebo | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Semaglutide 0.8 mg | Semaglutide 0.8 mg (With Titration) | Semaglutide 1.6 mg (With Titration) | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 47 | 43 | 48 | 42 | 43 | 47 | 45 | 50
Billion cells/litre (10^9/L) | 0.1 (1.7) | 0.0 (1.3) | -0.1 (1.4) | 0.3 (1.3) | -0.1 (1.6) | 0.5 (1.1) | 0.5 (1.4) | 0.3 (1.0) | 0.3 (1.4)

15. Secondary Outcome: Change From Baseline in Standard Safety Laboratory Parameter (Haematology; Thrombocytes)
Description: Change from baseline in thrombocytes was evaluated after 12 weeks of treatment. Post baseline (week 0) missing values were replaced using the LOCF approach.
Time Frame: Week 0, week 12
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Billion cells/litre (10^9/L)
Arm/Group | Placebo | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Semaglutide 0.8 mg | Semaglutide 0.8 mg (With Titration) | Semaglutide 1.6 mg (With Titration) | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 47 | 43 | 48 | 42 | 43 | 47 | 45 | 50
Billion cells/litre (10^9/L) | 9.0 (35.5) | 16.1 (30.2) | 10.8 (38.4) | 10.7 (47.9) | 5.4 (30.7) | 5.5 (50.6) | 15.9 (51.9) | 10.1 (37.1) | 16.7 (41.9)

16. Secondary Outcome: Change From Baseline in Standard Safety Laboratory Parameter (Haematology; Erythrocytes)
Description: Change from baseline in erythrocytes was evaluated after 12 weeks of treatment. Post baseline (week 0) missing values were replaced using the LOCF approach.
Time Frame: Week 0, week 12
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Trillion cells/litre (10^12/L)
Arm/Group | Placebo | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Semaglutide 0.8 mg | Semaglutide 0.8 mg (With Titration) | Semaglutide 1.6 mg (With Titration) | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 47 | 43 | 48 | 42 | 43 | 47 | 45 | 50
Trillion cells/litre (10^12/L) | -0.04 (0.21) | -0.06 (0.21) | -0.03 (0.31) | 0.08 (0.32) | -0.05 (0.25) | 0.03 (0.24) | 0.04 (0.24) | 0.04 (0.23) | 0.02 (0.38)

17. Secondary Outcome: Change From Baseline in Standard Safety Laboratory Parameter (Haematology; Leukocytes)
Description: Change from baseline in leukocytes was evaluated after 12 weeks of treatment. Post baseline (week 0) missing values were replaced using the LOCF approach.
Time Frame: Week 0, week 12
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Billion cells/litre (10^9/L)
Arm/Group | Placebo | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Semaglutide 0.8 mg | Semaglutide 0.8 mg (With Titration) | Semaglutide 1.6 mg (With Titration) | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 47 | 43 | 48 | 42 | 43 | 47 | 45 | 50
Billion cells/litre (10^9/L) | 0.05 (2.00) | 0.04 (1.39) | -0.16 (1.46) | 0.59 (1.50) | 0.14 (1.78) | 0.41 (1.44) | 0.70 (1.64) | 0.40 (1.15) | 0.26 (1.59)

18. Secondary Outcome: Change From Baseline in Standard Safety Laboratory Parameter (Biochemistry; Albumin)
Description: Change from baseline in albumin was evaluated after 12 weeks of treatment. Post baseline (week 0) missing values were replaced using the LOCF approach.
Time Frame: Week 0, week 12.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Placebo | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Semaglutide 0.8 mg | Semaglutide 0.8 mg (With Titration) | Semaglutide 1.6 mg (With Titration) | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 47 | 43 | 48 | 42 | 43 | 47 | 45 | 50
g/L | 0.402 (2.188) | 0.130 (2.505) | -0.091 (1.700) | -0.177 (2.331) | 0.303 (2.207) | 0.607 (2.034) | 0.271 (2.586) | 0.916 (1.933) | 0.846 (2.097)

19. Secondary Outcome: Change From Baseline in Standard Safety Laboratory Parameter (Biochemistry; Alkaline Phosphatase)
Description: Change from baseline in alkaline phosphatase was evaluated after 12 weeks of treatment. Post baseline (week 0) missing values were replaced using the LOCF approach.
Time Frame: Week 0, week 12.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Semaglutide 0.8 mg | Semaglutide 0.8 mg (With Titration) | Semaglutide 1.6 mg (With Titration) | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 47 | 43 | 48 | 42 | 43 | 47 | 45 | 50
U/L | -0.52 (8.78) | -1.66 (14.11) | -2.37 (11.87) | -2.35 (9.87) | -1.39 (12.24) | -2.81 (7.09) | -3.98 (9.02) | -1.89 (12.24) | -4.25 (10.90)

20. Secondary Outcome: Change From Baseline in Standard Safety Laboratory Parameter (Biochemistry; AST)
Description: Change from baseline in aspartate aminotransferase (AST) was evaluated after 12 weeks of treatment. Post baseline (week 0) missing values were replaced using the LOCF approach.
Time Frame: Week 0, week 12.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Semaglutide 0.8 mg | Semaglutide 0.8 mg (With Titration) | Semaglutide 1.6 mg (With Titration) | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 47 | 43 | 48 | 42 | 43 | 47 | 45 | 50
U/L | -1.09 (5.80) | 1.23 (8.93) | 0.24 (6.55) | -1.81 (9.54) | -0.37 (4.75) | -2.60 (7.38) | -4.07 (8.13) | -0.16 (6.12) | -2.13 (13.48)

21. Secondary Outcome: Change From Baseline in Standard Safety Laboratory Parameter (Biochemistry; ALAT)
Description: Change from baseline in alanine aminotransferase (ALAT) was evaluated after 12 weeks of treatment. Post baseline (week 0) missing values were replaced using the LOCF approach.
Time Frame: Week 0, week 12.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Semaglutide 0.8 mg | Semaglutide 0.8 mg (With Titration) | Semaglutide 1.6 mg (With Titration) | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 47 | 43 | 48 | 42 | 43 | 47 | 45 | 50
U/L | -2.41 (11.49) | 0.83 (8.23) | 0.68 (10.38) | -4.21 (15.15) | -2.13 (12.48) | -6.19 (12.26) | -6.55 (12.05) | -0.88 (8.96) | -1.83 (10.42)

22. Secondary Outcome: Change From Baseline in Standard Safety Laboratory Parameter (Biochemistry; Total Bilirubin)
Description: Change from baseline in total bilirubin was evaluated after 12 weeks of treatment. Post baseline (week 0) missing values were replaced using the LOCF approach.
Time Frame: Week 0, week 12.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Placebo | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Semaglutide 0.8 mg | Semaglutide 0.8 mg (With Titration) | Semaglutide 1.6 mg (With Titration) | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 47 | 43 | 48 | 42 | 43 | 47 | 45 | 50
umol/L | 0.7 (3.6) | -0.4 (2.8) | 0.6 (4.4) | 0.8 (3.7) | 0.7 (3.3) | 1.3 (5.4) | 0.4 (3.8) | -0.5 (4.7) | 0.2 (3.6)

23. Secondary Outcome: Change From Baseline in Standard Safety Laboratory Parameter (Biochemistry; Calcium, Total)
Description: Change from baseline in calcium, total was evaluated after 12 weeks of treatment. Post baseline (week 0) missing values were replaced using the LOCF approach.
Time Frame: Week 0, week 12.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Semaglutide 0.8 mg | Semaglutide 0.8 mg (With Titration) | Semaglutide 1.6 mg (With Titration) | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 47 | 43 | 48 | 42 | 43 | 47 | 45 | 50
mmol/L | 0.0 (0.1) | -0.0 (0.1) | -0.0 (0.1) | -0.0 (0.1) | 0.0 (0.1) | 0.0 (0.1) | -0.0 (0.1) | -0.0 (0.1) | 0.0 (0.2)

24. Secondary Outcome: Change From Baseline in Standard Safety Laboratory Parameter (Biochemistry; Calcium, Ionised)
Description: Change from baseline in calcium, ionised was evaluated after 12 weeks of treatment. Post baseline (week 0) missing values were replaced using the LOCF approach.
Time Frame: Week 0, week 12.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Semaglutide 0.8 mg | Semaglutide 0.8 mg (With Titration) | Semaglutide 1.6 mg (With Titration) | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 47 | 43 | 48 | 42 | 43 | 47 | 45 | 50
mmol/L | 0.00 (0.09) | -0.01 (0.11) | -0.04 (0.14) | -0.01 (0.07) | -0.01 (0.13) | 0.01 (0.09) | -0.02 (0.13) | -0.02 (0.11) | -0.01 (0.14)

25. Secondary Outcome: Change From Baseline in Standard Safety Laboratory Parameter (Biochemistry; Creatinine)
Description: Change from baseline in creatinine was evaluated after 12 weeks of treatment. Post baseline (week 0) missing values were replaced using the LOCF approach.
Time Frame: Week 0, week 12.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Placebo | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Semaglutide 0.8 mg | Semaglutide 0.8 mg (With Titration) | Semaglutide 1.6 mg (With Titration) | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 47 | 43 | 48 | 42 | 43 | 47 | 45 | 50
umol/L | -1.02 (7.206) | 0.936 (6.291) | -0.349 (11.22) | -2.31 (8.866) | -0.658 (11.08) | -1.67 (9.511) | 2.089 (7.099) | 0.841 (11.21) | -0.917 (6.270)

26. Secondary Outcome: Change From Baseline in Standard Safety Laboratory Parameter (Biochemistry; Potassium)
Description: Change from baseline in potassium was evaluated after 12 weeks of treatment. Post baseline (week 0) missing values were replaced using the LOCF approach.
Time Frame: Week 0, week 12.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Semaglutide 0.8 mg | Semaglutide 0.8 mg (With Titration) | Semaglutide 1.6 mg (With Titration) | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 47 | 43 | 48 | 42 | 43 | 47 | 45 | 50
mmol/L | 0.07 (0.37) | 0.08 (0.57) | 0.06 (0.42) | -0.02 (0.44) | 0.04 (0.61) | -0.02 (0.48) | -0.07 (0.46) | 0.10 (0.50) | -0.12 (0.47)

27. Secondary Outcome: Change From Baseline in Standard Safety Laboratory Parameter (Biochemistry; Sodium)
Description: Change from baseline in sodium was evaluated after 12 weeks of treatment. Post baseline (week 0) missing values were replaced using the LOCF approach.
Time Frame: Week 0, week 12.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Semaglutide 0.8 mg | Semaglutide 0.8 mg (With Titration) | Semaglutide 1.6 mg (With Titration) | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 47 | 43 | 48 | 42 | 43 | 47 | 45 | 50
mmol/L | 0.1 (2.3) | 0.0 (1.7) | -0.1 (2.6) | -0.1 (2.7) | 0.4 (2.4) | 0.2 (2.7) | 0.5 (2.7) | 0.7 (2.8) | 0.6 (2.3)

28. Secondary Outcome: Change From Baseline in Standard Safety Laboratory Parameter (Biochemistry; Urea)
Description: Change from baseline in urea was evaluated after 12 weeks of treatment. Post baseline (week 0) missing values were replaced using the LOCF approach.
Time Frame: Week 0, week 12.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Semaglutide 0.8 mg | Semaglutide 0.8 mg (With Titration) | Semaglutide 1.6 mg (With Titration) | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 47 | 43 | 48 | 42 | 43 | 47 | 45 | 50
mmol/L | -0.1 (1.2) | 0.1 (1.4) | -0.1 (1.3) | -0.4 (1.3) | -0.3 (1.6) | -0.5 (1.3) | -0.5 (1.3) | -0.1 (1.3) | -0.4 (1.1)

29. Secondary Outcome: Change From Baseline in Standard Safety Laboratory Parameter (Urinalysis; Glucose)
Description: Change from baseline in urine-glucose was measured in terms of number of subjects in each category (negative, positive, >=55 mmol/L, or missing) at week 0 and week 12 (i.e., change in each category in terms of number of subjects from week 0 to week 12).
Time Frame: Week 0, week 12
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Semaglutide 0.8 mg | Semaglutide 0.8 mg (With Titration) | Semaglutide 1.6 mg (With Titration) | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 47 | 43 | 48 | 42 | 43 | 47 | 45 | 50
Participants
  Week 0: Negative: number analyzed (Participants) | 46 | 47 | 43 | 48 | 41 | 43 | 47 | 45 | 50
  Week 0: Negative | 31 | 26 | 23 | 35 | 23 | 28 | 32 | 30 | 22
  Week 0: Positive: number analyzed (Participants) | 46 | 47 | 43 | 48 | 41 | 43 | 47 | 45 | 50
  Week 0: Positive | 13 | 18 | 15 | 11 | 15 | 10 | 12 | 10 | 20
  Week 0: >=55 mmol/L: number analyzed (Participants) | 46 | 47 | 43 | 48 | 41 | 43 | 47 | 45 | 50
  Week 0: >=55 mmol/L | 1 | 3 | 5 | 2 | 3 | 3 | 2 | 3 | 5
  Week 0: Missing: number analyzed (Participants) | 46 | 47 | 43 | 48 | 41 | 43 | 47 | 45 | 50
  Week 0: Missing | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 3
  Week 12: Negative: number analyzed (Participants) | 44 | 46 | 41 | 45 | 37 | 41 | 43 | 43 | 47
  Week 12: Negative | 34 | 28 | 28 | 35 | 30 | 39 | 39 | 35 | 39
  Week 12: Positive: number analyzed (Participants) | 44 | 46 | 41 | 45 | 37 | 41 | 43 | 43 | 47
  Week 12: Positive | 8 | 15 | 8 | 8 | 2 | 1 | 3 | 7 | 6
  Week 12: >=55 mmol/L: number analyzed (Participants) | 44 | 46 | 41 | 45 | 37 | 41 | 43 | 43 | 47
  Week 12: >=55 mmol/L | 2 | 2 | 3 | 1 | 2 | 0 | 0 | 1 | 0
  Week 12: Missing: number analyzed (Participants) | 44 | 46 | 41 | 45 | 37 | 41 | 43 | 43 | 47
  Week 12: Missing | 0 | 1 | 2 | 1 | 3 | 1 | 1 | 0 | 2

30. Secondary Outcome: Change From Baseline in Standard Safety Laboratory Parameter (Urinalysis; Haemoglobin)
Description: Change from baseline in urine-haemoglobin was measured in terms of number of subjects in each category (negative, trace, small, moderate/large and missing) at week 0 and week 12 (i.e., change in each category in terms of number of subjects from week 0 to week 12).
Time Frame: Week 0, week 12
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Semaglutide 0.8 mg | Semaglutide 0.8 mg (With Titration) | Semaglutide 1.6 mg (With Titration) | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 47 | 43 | 48 | 42 | 43 | 47 | 45 | 50
Participants
  Week 0: Negative: number analyzed (Participants) | 46 | 47 | 43 | 48 | 41 | 43 | 47 | 45 | 50
  Week 0: Negative | 45 | 45 | 41 | 45 | 38 | 39 | 43 | 43 | 45
  Week 0: Trace: number analyzed (Participants) | 46 | 47 | 43 | 48 | 41 | 43 | 47 | 45 | 50
  Week 0: Trace | 0 | 2 | 1 | 1 | 2 | 1 | 2 | 0 | 1
  Week 0: Small: number analyzed (Participants) | 46 | 47 | 43 | 48 | 41 | 43 | 47 | 45 | 50
  Week 0: Small | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1
  Week 0: Moderate: number analyzed (Participants) | 46 | 47 | 43 | 48 | 41 | 43 | 47 | 45 | 50
  Week 0: Moderate | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
  Week 0: Missing: number analyzed (Participants) | 46 | 47 | 43 | 48 | 41 | 43 | 47 | 45 | 50
  Week 0: Missing | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 3
  Week 12: Negative: number analyzed (Participants) | 44 | 46 | 41 | 45 | 37 | 41 | 43 | 43 | 47
  Week 12: Negative | 42 | 45 | 38 | 42 | 30 | 38 | 39 | 43 | 44
  Week 12: Trace: number analyzed (Participants) | 44 | 46 | 41 | 45 | 37 | 41 | 43 | 43 | 47
  Week 12: Trace | 0 | 0 | 1 | 2 | 1 | 1 | 2 | 0 | 1
  Week 12: Small: number analyzed (Participants) | 44 | 46 | 41 | 45 | 37 | 41 | 43 | 43 | 47
  Week 12: Small | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
  Week 12: Large: number analyzed (Participants) | 44 | 46 | 41 | 45 | 37 | 41 | 43 | 43 | 47
  Week 12: Large | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  Week 12: Missing: number analyzed (Participants) | 44 | 46 | 41 | 45 | 37 | 41 | 43 | 43 | 47
  Week 12: Missing | 0 | 1 | 2 | 1 | 3 | 1 | 1 | 0 | 2

31. Secondary Outcome: Change From Baseline in Standard Safety Laboratory Parameter (Urinalysis; Ketones)
Description: Change from baseline in urine-ketone was measured in terms of number of subjects in each category (negative, positive, >=55 mmol/L and missing) at week 0 and week 12 (i.e., change in each category in terms of number of subjects from week 0 to week 12).
Time Frame: Week 0, week 12
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Semaglutide 0.8 mg | Semaglutide 0.8 mg (With Titration) | Semaglutide 1.6 mg (With Titration) | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 47 | 43 | 48 | 42 | 43 | 47 | 45 | 50
Participants
  Week 0: Negative: number analyzed (Participants) | 46 | 47 | 43 | 48 | 41 | 43 | 47 | 45 | 50
  Week 0: Negative | 45 | 47 | 39 | 46 | 41 | 41 | 45 | 42 | 46
  Week 0: Positive: number analyzed (Participants) | 46 | 47 | 43 | 48 | 41 | 43 | 47 | 45 | 50
  Week 0: Positive | 0 | 0 | 4 | 2 | 0 | 0 | 1 | 1 | 1
  Week 0: Missing: number analyzed (Participants) | 46 | 47 | 43 | 48 | 41 | 43 | 47 | 45 | 50
  Week 0: Missing | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 3
  Week 12: Negative: number analyzed (Participants) | 44 | 46 | 41 | 45 | 37 | 41 | 43 | 43 | 47
  Week 12: Negative | 43 | 44 | 35 | 44 | 34 | 40 | 38 | 41 | 43
  Week 12: Positive: number analyzed (Participants) | 44 | 46 | 41 | 45 | 37 | 41 | 43 | 43 | 47
  Week 12: Positive | 1 | 1 | 4 | 0 | 0 | 0 | 4 | 2 | 2
  Week 12: Missing: number analyzed (Participants) | 44 | 46 | 41 | 45 | 37 | 41 | 43 | 43 | 47
  Week 12: Missing | 0 | 1 | 2 | 1 | 3 | 1 | 1 | 0 | 2

32. Secondary Outcome: Change From Baseline in Standard Safety Laboratory Parameter (Urinalysis; pH)
Description: Change from baseline in urine-pH was measured in terms of number of subjects in each category (pH=6.0, 6.5, 7.0, 7.5, 8.0, >=8.5 and missing) at week 0 and week 12 (i.e., change in each category in terms of number of subjects from week 0 to week 12).
Time Frame: Week 0, week 12
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Semaglutide 0.8 mg | Semaglutide 0.8 mg (With Titration) | Semaglutide 1.6 mg (With Titration) | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 47 | 43 | 48 | 42 | 43 | 47 | 45 | 50
Participants
  Week 0: 6.0: number analyzed (Participants) | 46 | 47 | 43 | 48 | 41 | 43 | 47 | 45 | 50
  Week 0: 6.0 | 16 | 13 | 19 | 11 | 10 | 11 | 14 | 8 | 12
  Week 0: 6.5: number analyzed (Participants) | 46 | 47 | 43 | 48 | 41 | 43 | 47 | 45 | 50
  Week 0: 6.5 | 13 | 18 | 15 | 21 | 13 | 13 | 10 | 16 | 11
  Week 0: 7.0: number analyzed (Participants) | 46 | 47 | 43 | 48 | 41 | 43 | 47 | 45 | 50
  Week 0: 7.0 | 11 | 12 | 8 | 10 | 12 | 8 | 12 | 14 | 19
  Week 0: 7.5: number analyzed (Participants) | 46 | 47 | 43 | 48 | 41 | 43 | 47 | 45 | 50
  Week 0: 7.5 | 4 | 3 | 0 | 5 | 5 | 8 | 7 | 3 | 2
  Week 0: 8.0: number analyzed (Participants) | 46 | 47 | 43 | 48 | 41 | 43 | 47 | 45 | 50
  Week 0: 8.0 | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 2 | 1
  Week 0: >=8.5: number analyzed (Participants) | 46 | 47 | 43 | 48 | 41 | 43 | 47 | 45 | 50
  Week 0: >=8.5 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2
  Week 0: Missing: number analyzed (Participants) | 46 | 47 | 43 | 48 | 41 | 43 | 47 | 45 | 50
  Week 0: Missing | 1 | 0 | 0 | 0 | 1 | 2 | 1 | 2 | 3
  Week 12: 6.0: number analyzed (Participants) | 44 | 46 | 41 | 45 | 37 | 41 | 43 | 43 | 47
  Week 12: 6.0 | 11 | 14 | 19 | 9 | 10 | 8 | 13 | 9 | 10
  Week 12: 6.5: number analyzed (Participants) | 44 | 46 | 41 | 45 | 37 | 41 | 43 | 43 | 47
  Week 12: 6.5 | 15 | 14 | 9 | 14 | 7 | 10 | 11 | 13 | 14
  Week 12: 7.0: number analyzed (Participants) | 44 | 46 | 41 | 45 | 37 | 41 | 43 | 43 | 47
  Week 12: 7.0 | 15 | 13 | 6 | 11 | 11 | 15 | 10 | 16 | 15
  Week 12: 7.5: number analyzed (Participants) | 44 | 46 | 41 | 45 | 37 | 41 | 43 | 43 | 47
  Week 12: 7.5 | 3 | 2 | 4 | 7 | 3 | 5 | 5 | 4 | 3
  Week 12: 8.0: number analyzed (Participants) | 44 | 46 | 41 | 45 | 37 | 41 | 43 | 43 | 47
  Week 12: 8.0 | 0 | 1 | 1 | 2 | 2 | 1 | 1 | 0 | 2
  Week 12: >=8.5: number analyzed (Participants) | 44 | 46 | 41 | 45 | 37 | 41 | 43 | 43 | 47
  Week 12: >=8.5 | 0 | 1 | 0 | 1 | 1 | 1 | 2 | 1 | 1
  Week 12: Missing: number analyzed (Participants) | 44 | 46 | 41 | 45 | 37 | 41 | 43 | 43 | 47
  Week 12: Missing | 0 | 1 | 2 | 1 | 3 | 1 | 1 | 0 | 2

33. Secondary Outcome: Change From Baseline in Standard Safety Laboratory Parameter (Urinalysis; Protein)
Description: Change from baseline in urine-protein was measured in terms of number of subjects in each category at week 0 (negative, 0.3 g/L, 1.0 g/L and missing) and week 12 (negative, trace, 0.3 g/L, 1.0 g/L, >=3.0 g/L and missing). i.e., change in each category in terms of number of subjects from week 0 to week 12.
Time Frame: Week 0, week 12
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Semaglutide 0.8 mg | Semaglutide 0.8 mg (With Titration) | Semaglutide 1.6 mg (With Titration) | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 47 | 43 | 48 | 42 | 43 | 47 | 45 | 50
Participants
  Week 0: Negative: number analyzed (Participants) | 46 | 47 | 43 | 48 | 41 | 43 | 47 | 45 | 50
  Week 0: Negative | 45 | 47 | 41 | 44 | 39 | 40 | 46 | 41 | 45
  Week 0: 0.3: number analyzed (Participants) | 46 | 47 | 43 | 48 | 41 | 43 | 47 | 45 | 50
  Week 0: 0.3 | 0 | 0 | 2 | 4 | 2 | 0 | 0 | 2 | 1
  Week 0: 1.0: number analyzed (Participants) | 46 | 47 | 43 | 48 | 41 | 43 | 47 | 45 | 50
  Week 0: 1.0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Week 0: Missing: number analyzed (Participants) | 46 | 47 | 43 | 48 | 41 | 43 | 47 | 45 | 50
  Week 0: Missing | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 3
  Week 12: Negative: number analyzed (Participants) | 44 | 46 | 41 | 45 | 37 | 41 | 43 | 43 | 47
  Week 12: Negative | 40 | 43 | 35 | 41 | 31 | 36 | 39 | 40 | 41
  Week 12: Trace: number analyzed (Participants) | 44 | 46 | 41 | 45 | 37 | 41 | 43 | 43 | 47
  Week 12: Trace | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Week 12: 0.3: number analyzed (Participants) | 44 | 46 | 41 | 45 | 37 | 41 | 43 | 43 | 47
  Week 12: 0.3 | 4 | 2 | 3 | 3 | 3 | 3 | 2 | 1 | 3
  Week 12: 1.0: number analyzed (Participants) | 44 | 46 | 41 | 45 | 37 | 41 | 43 | 43 | 47
  Week 12: 1.0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1
  Week 12: >=3.0: number analyzed (Participants) | 44 | 46 | 41 | 45 | 37 | 41 | 43 | 43 | 47
  Week 12: >=3.0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Week 12: Missing: number analyzed (Participants) | 44 | 46 | 41 | 45 | 37 | 41 | 43 | 43 | 47
  Week 12: Missing | 0 | 1 | 2 | 1 | 3 | 1 | 1 | 0 | 2

34. Secondary Outcome: Change From Baseline in Calcitonin
Description: Change from baseline in calcitonin was evaluated after 12 weeks of treatment. Post baseline (week 0) missing values were replaced using the LOCF approach.
Time Frame: Week 0, week 12.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Placebo | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Semaglutide 0.8 mg | Semaglutide 0.8 mg (With Titration) | Semaglutide 1.6 mg (With Titration) | Liraglutide 1.2 mg | Liraglutide 1.8 mg
Number analyzed (Participants) | 46 | 47 | 43 | 48 | 42 | 43 | 47 | 45 | 50
ng/L | 0.43 (1.85) | 0.48 (1.82) | -0.48 (4.29) | 0.62 (1.68) | 0.45 (1.79) | 0.87 (1.56) | 0.76 (1.78) | 0.55 (2.66) | 0.01 (2.07)

35. Secondary Outcome: Percentage of Subjects Developing Anti-semaglutide Antibodies
Description: Antibodies were measured after 12-week of treatment at week 17; percentage of participants with positive anti-semaglutide antibodies are presented here. Assessments of antibodies were not done for subjects allocated to the open-label liraglutide treatment arms.
Time Frame: After 12 weeks of treatment
Population: as for baseline characteristics
Measure: Number; unit: Percentage (%) of participants
Arm/Group | Placebo | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Semaglutide 0.8 mg | Semaglutide 0.8 mg (With Titration) | Semaglutide 1.6 mg (With Titration)
Number analyzed (Participants) | 46 | 47 | 43 | 48 | 42 | 43 | 47
Percentage (%) of participants | 0 | 0 | 0 | 0 | 0 | 0 | 3

ADVERSE EVENTS:
Time Frame: The results for adverse event presented here are treatment emergent, i.e., TEAE. A TEAE was defined as an event that had onset on or after the first date (week 0) on trial product and no later than 5 weeks after the last date on trial product (week 17), or that had onset before the first date on trial product and increases in severity during the treatment period until 5 weeks after the last date on trial product.
Description: The results are based on the safety analysis set, which included all randomised subjects who were exposed to at least 1 dose of trial product. 2 subjects randomised to semaglutide 0.8mg were mistakenly titrated, so actual treatment was semaglutide 0.8mg T. 2 subjects randomised to semaglutide 0.8mg T were mistakenly titrated to 1.6mg T, so actual treatment was semaglutide 1.6mg T.
Groups:
- Semaglutide 0.8 mg (With Titration): Subjects followed a 1-week titration period (semaglutide 0.4 mg once-weekly at week 1), followed by an 11-week treatment period of fixed doses semaglutide 0.8 mg, once-weekly. Semaglutide was injected s.c. in the abdomen, thigh or upper arm by using the NordiPen® on the same day of the week at a convenient time for the subjects. Semaglutide was given in adjunct to previous metformin therapy on a stable dose (minimum 1.5 g daily) or as monotherapy in case the diabetes was controlled by diet and exercise alone.
Arm/Group | Placebo | Semaglutide 0.1 mg | Semaglutide 0.2 mg | Semaglutide 0.4 mg | Semaglutide 0.8 mg | Semaglutide 0.8 mg (With Titration) | Semaglutide 1.6 mg (With Titration) | Liraglutide 1.2 mg | Liraglutide 1.8 mg
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/47 | 0/43 | 0/48 | 0/42 | 0/43 | 0/47 | 0/45 | 0/50
Serious Adverse Events (participants affected / at risk) | 1/46 | 1/47 | 1/43 | 2/48 | 0/42 | 1/43 | 2/47 | 0/45 | 0/50
Other Adverse Events (participants affected / at risk) | 9/46 | 23/47 | 14/43 | 27/48 | 32/42 | 29/43 | 39/47 | 18/45 | 21/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=46) | Semaglutide 0.1 mg (N=47) | Semaglutide 0.2 mg (N=43) | Semaglutide 0.4 mg (N=48) | Semaglutide 0.8 mg (N=42) | Semaglutide 0.8 mg (With Titration) (N=43) | Semaglutide 1.6 mg (With Titration) (N=47) | Liraglutide 1.2 mg (N=45) | Liraglutide 1.8 mg (N=50)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=46) | Semaglutide 0.1 mg (N=47) | Semaglutide 0.2 mg (N=43) | Semaglutide 0.4 mg (N=48) | Semaglutide 0.8 mg (N=42) | Semaglutide 0.8 mg (With Titration) (N=43) | Semaglutide 1.6 mg (With Titration) (N=47) | Liraglutide 1.2 mg (N=45) | Liraglutide 1.8 mg (N=50)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (5) | 3 (3) | 5 (6) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (5) | 1 (1) | 3 (8) | 3 (3) | 3 (4) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 2 (2) | 4 (4) | 10 (13) | 9 (10) | 23 (24) | 4 (4) | 6 (6)
Diabetic retinopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 5 (6) | 2 (3) | 7 (11) | 8 (12) | 7 (8) | 11 (14) | 2 (2) | 7 (9)
Dizziness (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (2) | 5 (5) | 0 (0) | 4 (6) | 4 (6) | 4 (7) | 6 (8) | 5 (6) | 4 (6)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (9) | 0 (0) | 0 (0) | 6 (22) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (4)
Headache (Nervous system disorders) | 3 (3) | 7 (11) | 3 (3) | 4 (10) | 5 (11) | 1 (2) | 3 (5) | 4 (8) | 2 (2)
Hypertension (Vascular disorders) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (4) | 6 (7) | 0 (0) | 4 (6) | 2 (3) | 2 (2) | 3 (4) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 4 (4) | 5 (8) | 13 (18) | 25 (38) | 17 (46) | 27 (61) | 11 (14) | 4 (4)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (5) | 7 (10) | 17 (22) | 13 (20) | 13 (19) | 4 (5) | 6 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.